CLINICAL TRIAL: NCT03621943
Title: Umbilical Cord Milking in Non-Vigorous Infants Developmental Followup (MINVIFU)
Acronym: MINVIFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director, Neonatal Research Institute, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MINVIFU
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Neurodevelopmental Abnormality
Keywords: Neurodevelopmental outcomes; Disability; Umbilical cord milking; Early cord clamping; Non-vigorous infants; Term infants; Near-Term infants; Developmental screening; Early childhood
MeSH Terms: interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: Randomization assignment was determined at time of enrollment in the primary study (Umbilical Cord Milking in Nonvigorous Infants Study NCT:03631940). The primary study model was a cluster randomized crossover trial.
Who Masked: Outcomes Assessor
Masking Description: Neurodevelopmental providers will be blinded to the randomization of the toddler during the examination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical Cord Milking (Active Comparator): At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped.
  Interventions: Procedure: Umbilical Cord Milking
- Early Cord Clamping (Active Comparator): The umbilical cord is clamped as soon as possible and within 60 seconds of delivery.
  Interventions: Procedure: Early Cord Clamping

INTERVENTIONS:
Procedure: Umbilical Cord Milking — At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped.
  Arms: Umbilical Cord Milking
Procedure: Early Cord Clamping — The umbilical cord is clamped as soon as possible and within 60 seconds of delivery.
  Arms: Early Cord Clamping

SUMMARY:
A sub-study to evaluate longer-term developmental outcomes in non-vigorous term and near-term newborns who receive umbilical cord milking in comparison to those who undergo early cord clamping at delivery.

DETAILED DESCRIPTION:
This sub-study investigates the potential difference in neurodevelopmental outcomes during early childhood between newborns who undergo umbilical cord milking and those who experience early cord clamping at birth. The developmental progress of participants is evaluated using the Ages and Stages Questionnaire-3 which measures five developmental areas: communication, problem-solving, fine motor skills, gross motor skills, and personal-social behavior. Additionally, the Modified Checklist for Autism in Toddlers is employed as a secondary assessment. The recruitment of participants is conducted through the primary study Umbilical Cord Milking in Nonvigorous Infants trial (NCT03631940) with the method of umbilical cord management for each newborn being dictated by the randomized treatment allocation of the primary study.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the primary trial NCT:03631940 and parental written consent to participate in developmental follow-up through 2 years of age was obtained.
* Enrolled in the primary trial NCT:03631940 and did not survive to 2 years.

Exclusion Criteria:

- Enrolled in the primary trial NCT:03631940 but parent/guardian declined consent to developmental follow-up participation.

Ages: 22 Months to 26 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1207 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2023-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anup Katheria, MD, Principal Investigator — Neonatologist
Locations (10):
- United States (7):
  - University of California, Davis, Davis, California
  - Loma Linda Medical Center, Loma Linda, California
  - Sharp Grossmont Hospital, San Diego, California
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California
  - George Washington University, Washington D.C., District of Columbia
  - Providence St. Vincent Medical Center, Portland, Oregon
  - University of Utah/IMH, Salt Lake City, Utah
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Dalhousie University, Dalhousie, New Brunswick
- Poznan University of Medical Science, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study design: cluster crossover randomization of 10 maternity hospitals to perform cord milking or early cord clamping. Participants were recruited among non-vigorous newborn born during the initial study period: January 2019 - January 2020 and crossover period: February 2020 - March 2021.
Pre-assignment Details: Hospital sites were informed of their randomization status two months before initiation of recruitment to permit time for physician and staff education on the assigned intervention. Prior to the start of recruitment in the crossover study period a 1 to 2-month washout period for each hospital site was specified by the protocol for the purpose of site hospital staff education on the change in assigned intervention and to assess adherence prior to recruitment initiation in the second study period.
Units Other Than Participants: Hospital
Groups:
- Umbilical Cord Milking Then Early Cord Clamping Site Randomization - Infant: In the first study period infants assessed as non-vigorous at delivery had the umbilical cord is grasped by the obstetric provider, and blood was pushed toward the infant 4 times before the cord is clamped.
  In the second study period infants assessed as non-vigorous at delivery had the umbilical cord clamped by 60 seconds of life.
- Early Cord Clamping Then Umbilical Cord Milking Site Randomization - Infant: In the first study period infants assessed as non-vigorous at delivery had the umbilical cord clamped as soon as possible and within 60 seconds of delivery. In the second study period umbilical cord was grasped by the obstetric provider, and blood was pushed toward the infant 4 times before the cord is clamped.
Period: First Randomized Intervention
Arm/Group | Umbilical Cord Milking Then Early Cord Clamping Site Randomization - Infant | Early Cord Clamping Then Umbilical Cord Milking Site Randomization - Infant
Started | 284; 5 Hospital (Includes all infants whose parents provided consent for their participation in the developmental follow-up study. These participants delivered at a hospital randomized to perform umbilical cord milking on all non-vigorous infants delivered in the first study period.) | 321; 5 Hospital (Includes all infants whose parents provided consent for their participation in the developmental follow-up study. These participants delivered at a hospital randomized to perform early cord clamping on all non-vigorous infants delivered in the first study period.)
Completed | 230; 5 Hospital (Includes all children whose parents provided consent for participation in the developmental follow-up study in the first study period and whose caregiver completed the Ages and Stages 3rd edition questionnaire when the child reached 2 years of age.) | 264; 5 Hospital (Includes all children whose parents provided consent for participation in the developmental follow-up study in the first study period and whose caregiver completed the Ages and Stages 3rd edition questionnaire when the child reached 2 years of age.)
Not Completed | 54; 0 Hospital | 57; 0 Hospital
Not completed — Lost to Follow-up | 51 | 54
Not completed — Withdrawal by Subject | 3 | 3
Period: Crossover Randomized Intervention
Arm/Group | Umbilical Cord Milking Then Early Cord Clamping Site Randomization - Infant | Early Cord Clamping Then Umbilical Cord Milking Site Randomization - Infant
Started | 280; 5 Hospital (In this study design the participants recruited in the initial study period with treatment of umbilical cord milking did not continue on to the crossover period. In the cross over period hospital sites recruited new participants with a target enrollment equivalent to the site's recruitment in the initial study period and performed early cord clamping in the second study period.) | 322; 5 Hospital (Includes all infants whose parents provided consent for their participation in the developmental follow-up study. These participants delivered at a hospital randomized to perform umbilical cord milking on all non-vigorous infants delivered in the second study period.)
Completed | 205; 5 Hospital (Includes all children whose parents provided consent for participation in the developmental follow-up study in the second study period and whose caregiver completed the Ages and Stages 3rd edition questionnaire when the child reached 2 years of age.) | 272; 5 Hospital (Includes all children whose parents provided consent for participation in the developmental follow-up study in the second study period and whose caregiver completed the Ages and Stages 3rd edition questionnaire when the child reached 2 years of age.)
Not Completed | 75; 0 Hospital | 50; 0 Hospital
Not completed — Lost to Follow-up | 75 | 45
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for all infant participants whose caregiver provided consent to participation in the 2-year follow-up study and whose caregiver completed an ASQ-3 Questionnaire when the child reached 2 years of age. All presented counts represent unique participants.
Groups:
- Umbilical Cord Milking Treatment Only- Infant & Maternal Baseline Measures: Baseline measures presented by randomized treatment assignment. Includes all infants who were assigned to umbilical cord milking (umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped) treatment based on hospital randomization. Maternal data is presented for all participating mothers. Only unique participants are presented.
- Early Cord Clamping Treatment Only- Infant & Maternal Baseline Measures: Baseline measures presented by randomized treatment assignment. Includes all infants who were assigned to the early cord clamping (The umbilical cord is clamped as soon as possible and within 60 seconds of delivery) treatment at delivery based on hospital randomization. Maternal data is presented for all participating mothers. Only unique participants are presented.
- Total: Total of all reporting groups
Arm/Group | Umbilical Cord Milking Treatment Only- Infant & Maternal Baseline Measures | Early Cord Clamping Treatment Only- Infant & Maternal Baseline Measures | Total
Number analyzed (Participants) | 502 | 469 | 971
Age, Continuous [Median (Inter-Quartile Range); unit: weeks] — Infant's gestational age at delivery
  weeks
    Infant's gestational age at birth | 39 [38 to 40] | 39 [38 to 40] | 39 [38 to 40]
Age, Customized [Mean (Standard Deviation); unit: years, maternal age at delivery] — Age of the mother at childbirth
  years, maternal age at delivery
    Maternal age at delivery | 31 (5) | 31 (6) | 31 (6)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of infant participants. Maternal sex was not collected as a variable in the study dataset.
  Participants
    Infant sex: Female | 224 | 201 | 425
    Infant sex: Male | 278 | 268 | 546
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of infant participants as reported by birth parents.
  Participants
    Infant Ethnicity: Hispanic or Latino | 100 | 102 | 202
    Infant Ethnicity: Not Hispanic or Latino | 375 | 302 | 677
    Infant Ethnicity: Unknown or Not Reported | 27 | 65 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of birth mother of participating infant as self-reported.
  Participants
    Maternal Ethnicity: Hispanic or Latino | 86 | 88 | 174
    Maternal Ethnicity: Not Hispanic or Latino | 393 | 321 | 714
    Maternal Ethnicity: Unknown or Not Reported | 23 | 60 | 83
Race (NIH/OMB) [Count of Participants; unit: Participants] — Infant race as reported by birth parents
  Participants
    Infant Race: American Indian or Alaska Native | 5 | 2 | 7
    Infant Race: Asian | 31 | 37 | 68
    Infant Race: Native Hawaiian or Other Pacific Islander | 2 | 5 | 7
    Infant Race: Black or African American | 29 | 29 | 58
    Infant Race: White | 287 | 260 | 547
    Infant Race: More than one race | 87 | 86 | 173
    Infant Race: Unknown or Not Reported | 61 | 50 | 111
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of birth mother of participating infant as self-reported.
  Participants
    Maternal Race: American Indian or Alaska Native | 12 | 5 | 17
    Maternal Race: Asian | 39 | 46 | 85
    Maternal Race: Native Hawaiian or Other Pacific Islander | 5 | 8 | 13
    Maternal Race: Black or African American | 35 | 36 | 71
    Maternal Race: White | 322 | 283 | 605
    Maternal Race: More than one race | 28 | 30 | 58
    Maternal Race: Unknown or Not Reported | 61 | 61 | 122
Region of Enrollment [Number; unit: infant participants]
  Canada | 159 | 159 | 318
  United States | 326 | 297 | 623
  Poland | 17 | 13 | 30
Number of neonates born to a mother with at least some college education [Number; unit: infant participants] — Baseline measure includes all infant-mother dyads who self-disclosed maternal highest level of education at the time of consent to long term follow-up participation. Population: Maternal level of education was not collected for infant-mother dyads who refused to self-disclose birth mother's highest level of education at time of consent to long-term follow-up. All participants represented are unique with no duplicate participants
  infant participants
    number analyzed (Participants) | 446 | 406 | 852
    (all) | 349 | 321 | 670
Count of newborns delivered by a mother with diabetes [Number; unit: number of infant participants] — Total number of infant participants whose mother had diabetes during gestation.
  number of infant participants | 72 | 63 | 135
Count of newborns delivered by a mother with hypertension [Number; unit: number of infant participants] — Total infant participants born to a mother with high blood pressure during gestation.
  number of infant participants | 89 | 81 | 170
Count of newborns delivered by a mother with intrauterine inflammation/infection [Number; unit: infant participants] — Total number of infants delivered by a mother with an intrauterine infection or inflammation condition during gestation.
  infant participants | 54 | 62 | 116
Count of newborns delivered by a mother with Group B Streptococcus [Number; unit: infant participants] — Total number of infants delivered by a mother with a positive Group B Streptococcus culture Population: One neonate-mother dyad in the umbilical cord clamping group has unknown screening status for Group B Streptococcus.
  infant participants
    number analyzed (Participants) | 501 | 469 | 970
    (all) | 114 | 88 | 202
Duration of fetal membrane rupture prior to delivery [Median (Inter-Quartile Range); unit: hours since amnionic sac rupture] | 6 [1 to 14] | 5 [1 to 14] | 6 [1 to 14]
Count of infants delivered by a mother administered narcotics/CNS depressants before delivery [Number; unit: infant participants] — Total count of infants delivered by a mother administered narcotics/central nervous system depressants within 2 hours of delivery.
  infant participants | 51 | 51 | 102
Count of infants delivered by cesarean section [Number; unit: infant participants] — Total number of infants born via surgical delivery (cesarean section)
  infant participants | 246 | 206 | 452
Count of infants born to a mother with a multiple birth pregnancy [Number; unit: infant participants] — Total number of infants that were part of a multiple gestation pregnancy. Population: Reported for all infant participants with maternal multiple gestation status collected.
  infant participants
    number analyzed (Participants) | 501 | 467 | 968
    (all) | 13 | 18 | 31
Count of newborns who were administered the correct randomized treatment at delivery [Number; unit: infant participants] — Total number of neonates who received the correct treatment assigned to the delivery hospital for all non-vigorous newborn delivered during the two enrollment periods.
  infant participants | 486 | 465 | 951

OUTCOME MEASURES:

1. Primary Outcome: Total and Domain Scores on the Ages and Stages Questionnaire, Third Edition.
Description: Neurodevelopmental Outcome at 2 Years of Age defined as overall and domain scores on the Ages and Stages, third edition. Questionnaire. Minimum score of 0 and maximum score of 60 per domain. Scores from 5 subscales are summed to obtain a total score. 5 domains assessed include communication, gross motor, fine motor, problem solving, personal social with a total minimum score of 0 and maximum score of 300. Higher scores indicate a lower risk of developmental delays or conditions
Time Frame: 22 to 26 months
Population: Children who had Ages and Stages, third edition. Questionnaire scores available at 2 years or died before age 2 years.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Umbilical Cord Milking - Infant: At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped.
- Early Cord Clamping - Infant: The umbilical cord is clamped as soon as possible and within 60 seconds of delivery.
Arm/Group | Umbilical Cord Milking - Infant | Early Cord Clamping - Infant
Number analyzed (Participants) | 502 | 469
score on a scale
  Communication score | 55 [40 to 60] | 55 [40 to 60]
  Gross motor score | 60 [50 to 60] | 60 [50 to 60]
  Fine motor score | 50 [45 to 60] | 50 [45 to 60]
  Problem solving score | 50 [40 to 55] | 50 [40 to 60]
  Personal-social score | 50 [40 to 55] | 50 [45 to 55]
  Total Ages and Stages Questionnaire score | 255 [225 to 280] | 255 [230 to 280]
Statistical Analysis 1: Comparison: Umbilical Cord Milking - Infant vs Early Cord Clamping - Infant; Total score on the Ages and Stages Questionnaire, 3rd ed; Test type: Superiority; p = 0.87, hierarchical generalized linear mixed mo; hierarchical generalized linear mixed models; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-6.36 to 5.37]

2. Secondary Outcome: Score Ranges on the Modified Checklist for Autism in Toddlers Questionnaire
Description: Modified Checklist for Autism in Toddlers. Minimum score of 0 and maximum score of 20. Higher scores indicate higher risk for autism spectrum disorder. Total scores of 0 to 2 indicates a low risk of autism spectrum disorder. Total scores of 3 to 7 indicates a moderate risk of autism spectrum disorder. Total scores of 8 to 20 indicate high risk of autism spectrum disorder.
Time Frame: 22-26 months
Population: Child participants with a total score from the Modified Checklist for Autism in Toddlers or died before the age of 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Milking - Infant | Early Cord Clamping - Infant
Number analyzed (Participants) | 486 | 441
Participants
  Score 0-2 | 441 | 404
  Score 3-7 | 34 | 31
  Score 8-20 | 11 | 6

ADVERSE EVENTS:
Time Frame: Infant's birth to 2 years of age.
Description: Adverse events were assessed for infant participants only and were collected from delivery to 2 years of age.
Arm/Group | Umbilical Cord Milking - Infant | Early Cord Clamping - Infant
All-Cause Mortality (participants affected / at risk) | 2/502 | 5/469
Serious Adverse Events (participants affected / at risk) | 0/502 | 0/469
Other Adverse Events (participants affected / at risk) | 0/502 | 0/469

LIMITATIONS AND CAVEATS:
This study was conducted in relatively high-income academic centers. Most women had sufficient prenatal care, and almost 80% of the mothers had some college education.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT03621943/Prot_SAP_000.pdf